CLINICAL TRIAL: NCT00245310
Title: Evaluation of the Indocyangreen Elimination as a Prognostic Marker in Decompensated Cirrhosis and Acute Liver Failure
Brief Title: Indocyangreen Elimination in Cirrhosis and Acute Liver Failure
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Other Study IDs: LiMON
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2010-10-11 (Estimated); Status verified 2008-11

CONDITIONS: Acute Liver Failure; Liver Cirrhosis
Keywords: ICG clearance; liver cirrhosis; acute liver failure; prognosis
MeSH Terms: conditions — Liver Failure, Acute; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Indocyangreen (ICG) clearance

SUMMARY:
Indocyangreen (ICG)is totally biliary eliminated and corresponds to hepatocyte function and liver perfusion.

The ICG-clearance will be evaluated as a prognostic marker in liver disease.

DETAILED DESCRIPTION:
patients with acute liver failure or advanced liver disease will be studied. ICG-clearance will be correlated with established clinical scores and outcome.

ELIGIBILITY:
Inclusion Criteria:

* acute liver failure OR end-stage liver disease
* normal hepatic perfusion by doppler ultrasound

Exclusion Criteria:

* portal vein thrombosis
* allergy to ICG or iodine
* thyroid disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2005-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Encke, PD Dr. med., Principal Investigator — Heidelberg University
Locations (1):
- University of Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Merle U, Sieg O, Stremmel W, Encke J, Eisenbach C. Sensitivity and specificity of plasma disappearance rate of indocyanine green as a prognostic indicator in acute liver failure. BMC Gastroenterol. 2009 Dec 3;9:91. doi: 10.1186/1471-230X-9-91. PMID 19954554